CLINICAL TRIAL: NCT01698151
Title: Prognosis and Treatment of COPD in Primary Care-use of Biomarkers
Acronym: PROTECCT-M
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government); Region of Southern Denmark (Other)
Responsible Party: Principal Investigator, Frans Boch Waldorff, Principal Investigator, University of Southern Denmark
Other Study IDs: S-20110163
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational study in primary care aiming to validate biomarkers for chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* 40 years old or more,
* diagnosis of COPD in primary care

Exclusion Criteria:

* Major psychiatric illness,
* inability to visit primary care doctor,
* inability to understand danish language,

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in primary care on the Fyn island, Denmark
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-10; Primary Completion 2016-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Hospitalization | December 1, 2015

CONTACTS AND LOCATIONS:
Overall Officials: Frans Boch Waldorff, MD, PhD, Principal Investigator — University of Southern Denmark
Locations (37):
- Denmark (37):
  - Nyhegn, Søndergaard, Trabjerg og Vilhelmsen, Middelfart, Fyn
  - Lægerne J.B. Winsløws Vej, Odense, Fyn
  - Peter Larsen, Odense, Fyn
  - Peer Kirkebjerg, Odense C, Fyn
  - Lægerne Lærkevej, Otterup, Fyn
  - Søndersø Lægehus, Søndersø, Fyn
  - Lægerne i Bullerup, Agedrup
  - Lægehuset Skelvænget, Assens
  - Lægerne i Nr. Lyndelse, Årslev
  - Aaruplægerne, Årup
  - Lægerne Lægehuset, Faaborg
  - Per Andersen, Faaborg
  - Lægehuset i Gislev, Gislev
  - Haarbylægerne, Haarby
  - Jordløselægerne, Haarby
  - Lægerne i Hesselager, Hesselager
  - Lægerne Glenthøj & Nielsen, Kerteminde
  - Lægerne Tronegaard-Madsen og Schmidt, Kerteminde
  - Muusgaarden, Kerteminde
  - Lægerne i Kværndrup, Kværndrup
  - Lægerne i Havnegade, Middelfart
  - Lægehuset i Morud, Morud
  - Lægerne Nr. Voldgade, Nyborg
  - Lægerne Nyenstad, Nyborg
  - Bylægen Peer Kirkebjerg & Speciallæge Nanna Kirkebjerg, Odense
  - Læge Bo Gamborg Nielsen, Odense
  - Annette Tornøe, Odense C
  - Kirsten Wengler, Odense C
  - Læge Thore Eriksen, Odense C
  - Lægerne Agertoft og Petersen, Odense C
  - Almen Medicinsk Lægeklinik, Odense SØ
  - Lægerne Banepladsen, Otterup
  - Lægerne i Østergade, Ringe
  - Lægehuset Rudkøbing I/S, Rudkøbing
  - Lægerne Ørstedsgade, Rudkøbing
  - Lægerne Toldbodvej, Svendborg
  - Lægehuset i Vissenbjerg, Vissenbjerg

REFERENCES:
- [Derived] Sondergaard J, Halling A. The PROTECCT-M study: a cohort study investigating associations between novel specific biomarkers, patient-related, healthcare system markers and the trajectory of COPD patients treated in primary care. BMC Pulm Med. 2014 May 20;14:88. doi: 10.1186/1471-2466-14-88. PMID 24886233